CLINICAL TRIAL: NCT06192121
Title: The Effect of Self-Care Disability Theory-Based Web-Based Education for Individuals With Type-2 Diabetes on Care Outcomes
Brief Title: Web-Based Education for Individuals With Type-2 Diabetes
Acronym: Type-2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Kemal Elyeli, Research Asistant, PhD (c), Near East University, Turkey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NearEastU1
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; Internet-Based Intervention; Models, Nursing; Randomised Control Trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Randomised Control Trial
Who Masked: Participant
Masking Description: Simple Randomization and single blinding will be done.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standart Health Care which is provided regular from ministry of health for 3 months
- Experiment (Experimental): Standart Health Care which is provided regular from ministry of health for 3 months Web Based Education for 3 months 3 reminder messages (SMS) per week
  Interventions: Other: Web Based Education

INTERVENTIONS:
Other: Web Based Education — In this research, a reminder message will be sent 3 times a week along with web-based training.
  Arms: Experiment

SUMMARY:
Type and Aim of Research This research will be conducted as a randomised controlled experimental study design to test the effect of web-based diabetes education on the quality of life and self-care activities of individuals with Type 2 Diabetes.

Place and Time of the Study This research will be conducted between September 2023 and March 2024 with individuals registered to the Cyprus Turkish Diabetes Association.

Population and Sample of the Study The population of the study consisted of individuals with Type-2 diabetes who applied to the Cyprus Turkish Diabetes Centre. The sample of the study included individuals with type-2 diabetes who met the inclusion criteria at the Turkish Cypriot Diabetes Centre.

Sample size was calculated using G Power statistical programme (n=74).

In order to evaluate the effectiveness in the experimental and control groups, simple randomisation was performed to ensure the similarity of the two groups. Randomisation was applied after the pre-tests.

The data of the study will be collected by Sociodemographic Data Form, Diabetes Specific Quality of Life Scale, Diabetes Self-Care Activities Questionnaire, Website Analysis and Measurement Inventory. The forms will be applied to the participants face to face.

People in the experimental group, whose information was sent to the researcher, will receive reminder messages twice a week (Wednesday-Friday) during the 3-month follow-up period via the website. No intervention will be applied to the control group. The post-test will be applied.

DETAILED DESCRIPTION:
The Effect of Self-Care Disability Theory-Based Web-Based Education for Individuals with Type-2 Diabetes on Care Outcomes

Purpose of the Study The aim of this study is to determine the effect of web-based diabetes education developed on the basis of self-care deficiency on individuals' quality of life and self-care activities.

Hypotheses of the Study

H0: There is no difference between the total mean score of the Diabetes Specific Quality of Life scale between the experimental and control groups of the Web-based diabetes education programme prepared on the basis of the Self-Care Disability Theory.

H0: There is no difference between the mean scores of the Diabetes Self-Care Activities scale between the experimental and control groups of the Web-based diabetes education programme prepared on the basis of the Self-Care Disability Theory.

METHOD

Type of Research This research will be conducted as a randomised controlled experimental study design to test the effect of web-based diabetes education on the quality of life and self-care activities of individuals with Type 2 Diabetes.

Place and Time of the Study This research will be conducted between September 2023 and March 2024 with individuals registered to the Cyprus Turkish Diabetes Association.

Population and Sample of the Study The population of the study consisted of individuals with Type-2 diabetes who applied to the Cyprus Turkish Diabetes Centre. The sample of the study included individuals with type-2 diabetes who met the inclusion criteria at the Turkish Cypriot Diabetes Centre.

Cyprus Turkish Diabetes Association The Cyprus Turkish Diabetes Association was established in Nicosia in 1994. The aim of the association is to improve the quality of life of diabetics and their relatives and to increase awareness of diabetes. Among the visions published by the association; freeing people from the restrictions of diabetes, providing the highest quality care and information to everyone, ending ignorance and discrimination, gaining an international understanding of diabetes and its organisations, and creating a world without diabetes.

Research Criteria

Inclusion Criteria

* Literate in Turkish,
* With access to the Internet,
* Diagnosed with Type II Diabetes,
* Mental competence,
* Individuals who volunteered to participate in the study were included.

Exclusion Criteria

* Cannot use a computer or smartphone,
* Under 18 years of age,
* With Type 1 Diabetes
* Working in the field of health and receiving health education in any field,
* Individuals who participated in the pre-application were not included in the study.

Calculation of Sample Size Sample size was calculated using G Power statistical programme. In order to reach the minimum and maximum sample numbers to be sampled, it is stated that the effect sizes of these studies should be determined from the mean and standard deviation levels of the intervention and control groups obtained from the scales obtained from previous, similar studies. The effect size of Wu, which is the closest study to our study, was found to be 0.70 in his study (n:145) conducted with the Diabetes Self-Care Activities Questionnaire in individuals with diabetes. As a result of the calculation made by taking 90% power and 0.05 error margin as well as the effect sizes obtained from the studies for the sample size, the sample number for each of the intervention and control groups for our study was determined as 36 individuals in each group according to the Diabetes Self-Care Activities Questionnaire with an effect size of 0.70. According to these results, a total of 72 patients (36 intervention and 36 control) should be included in the intervention and control groups. However, the sample was increased by 10% against the possibility of sample loss during the study, and the sample of the study was initially determined as a total of 80 patients, 40 intervention and 40 control.

Randomization In order to evaluate the effectiveness in the experimental and control groups, randomization was performed to ensure the similarity of the two groups. By choosing the simple randomization method, an equal number of samples (experiment: 40, control: 40) were provided for the experimental and control groups. After informed consent and pretests are completed, assignments to groups will be made by a different instructor in order to avoid bias. Assignment to groups will be done using the simple randomization method using the web program and the closed envelope method with a simple table of numbers. The group the individual will be in will be communicated to the researcher in a sealed envelope before the intervention.

Blinding Blinding will be done in data collection, statistics and reporting in the research. In the research, after obtaining pre-test data, randomization and data entry (pre- and post-tests and data transfer to the computer) will be carried out by a nursing faculty member other than the researcher who is unaware of the experimental and control groups. Data entries were entered with the code "A" and "B" without specifying the experimental or control group. Data analysis and writing of the research report will be coded as "A" and "B" groups. After the statistical analysis is performed and the research report is written, the coding for the experimental and control groups will be explained to the researcher by the coder.

Data Collection Tools Data of the research; It will be collected with the Sociodemographic Data Form, Diabetes-Specific Quality of Life Scale, Diabetes Self-Care Activities Survey, Website Analysis and Measurement Inventory. The forms will be administered to participants face to face.

Socio-demographic Data Form The socio-demographic questionnaire, prepared by the researchers after literature review, consists of 23 questions that determine the characteristics of individuals such as age, gender and educational status.

Diabetes-Specific Quality of Life Scale The Diabetes-Specific Quality of Life Scale, defined by Jacobson consists of four subscales and 46 items: psychological satisfaction with treatment, psychological impact, diabetes-related anxiety, and social/occupational anxiety. Each item in the scale is scored between 1-5 points. In the dimension of psychological satisfaction with the treatment (questions 22-24), the answer "very satisfied" is calculated as 1 point, the answer "very dissatisfied" is calculated as 5 points, while in the other dimensions the answer "never" is calculated as 1 point, and the answer "always" is calculated as 5 points. The total score of the scale varies between 46-230. The total scale score and each subscale score are divided by the number of items, and the scores of 1 are converted into 5 points to obtain the total scale score. According to the scale total scores, high scores indicate good quality of life. Subscale Cronbach's alpha values of the original scale are between 0.66 and 0.92, and the test-retest value is 0.78 and 0.92. A Turkish validity and reliability study of the scale was conducted by Yıldırım. The total Cronbach alpha value of the scale was found to be 0.89, and the Cronbach alpha values for the subscales were found to be between 0.80-0.94.

Diabetes Self-Care Activities Survey The Diabetes Self-Care Activities Questionnaire was developed by Toobert. In the survey, individuals; It is asked how many days (days/week) in the last seven days the patient performed self-care activities under the headings of diet, exercise, blood sugar test, foot care and smoking. The answers are marked as days (0-7) on a number line, and the 11th item, which only questions smoking, is stated as 0 - I do not smoke, 1 - I smoke (amount/piece of cigarettes smoked). Each subscale of the scale is scored separately and can be used independently.

The Turkish validity and reliability study of the scale was conducted by Coşansu.

Website Analysis and Measurement Inventory

Website Analysis and Measurement Inventory (WAMMI) is a scale based on usability and software evaluation for international software standards. WAMMI is used to evaluate web sites in many areas. It has translations in many European languages. The inventory measures attractiveness, controllability, It includes the sub-dimensions of efficiency, helpfulness, learnability and global usability. WAMMI scores are expressed as a percentage, the higher the percentage, the more useful the website is. The average score is calculated as the numerical average of the individual scores scored by the participants. Standard deviation, variability in the data A reasonable value for standard deviation for this type of data is 20. If all participants have a common opinion about website evaluations, the standard deviation is expected to be smaller. If participants have different opinions, the standard deviation is much larger, with a standard deviation above 30. deviation indicates that there are two or more groups of participants with very different opinions about the usability of the website.

Application of Research

During the implementation of the research, first of all, 181 people who applied to the Turkish Cypriot Diabetes Association were reached by the researcher. Among the 101 people reached; 76 people were not included in the study because they had type 1 diabetes, 14 people could not use a computer or smartphone, 4 people were healthcare workers, 3 people did not agree to participate in the research, and 4 people were not mentally competent (n: 80). As part of the pre-test, the sociodemographic questionnaire, diabetes-specific quality of life scale, and diabetes self-care activities scale were applied to the participants.

In order to carry out the randomization of the determined research sample, help was received from another researcher and the Simple Randomization Method was applied and the information of the individuals in the experimental (n: 40) and control (n: 40) groups was conveyed to the researcher.

The website was installed on the phones of the people in the experimental group, whose information was forwarded to the researcher.

During the 3-month follow-up period, reminder messages will be sent to individuals in the experimental group twice a week (Wednesday-Friday), while no intervention will be applied to the control group.

In order to prevent bias within the scope of the post-test, the post-test data of the participants will be obtained with the help of an expert researcher in the field, through appointments made at the Turkish Cypriot Diabetes Center. While the diabetes-specific quality of life scale and diabetes self-care activities survey will be applied to the control group, website analysis and measurement inventory will also be applied to the control group, unlike these surveys.

After the research is completed, the control group will be informed about the website and they will be able to benefit from the website.

Applications for Web-Based Training Program Development The training program development process, which was methodologically planned for the purpose of the research to develop a training program for individuals with Type 2 diabetes, is explained below.

Web designing

The following steps were followed during web design:

* Editing the topics and content of the website; Today's national and international websites, existing training booklets, current literature (meta-analyses, systematic reviews, original articles, books) and current guides used in this field were used.
* The content of the website is Public Health Nursing Lecturer (4 people), Internal Medicine Nursing Lecturer (1 person), Diabetes Education Nurses (1 person), Mental Health and Diseases Lecturer (2 people) and Dietetics and Nutrition Department Lecturer ( It was evaluated by 1 person) and edited with topic suggestions.
* The website is designed to be mobile compatible.
* Website: The website address is www.kibrisdiyabethemsireligi.com. The website has been prepared in parallel with the information provided in the literature and expert opinions; It is supported with videos, pictures, interactive forms, e-mail help and contact information.
* After the preparation of the website, it was evaluated by 5 researchers and 2 software experts who work in the field of web-based education.

Website Pre-Application

In order to test the understandability of the website for patients, a preliminary application was carried out at the Turkish Cypriot Diabetes Association between July and August 2023, for 10 individuals diagnosed with type 2 diabetes.

In the first interview with individuals who meet the research inclusion criteria and agree to participate in the research;

* As part of the pretest, the Sociodemographic Questionnaire, Diabetes-Specific Quality of Life Scale and Diabetes Self-Care Activities Survey were administered by the researcher.
* A username and password were created by the researcher to log in to the website.
* Participants were explained how to log in to the website by logging in with the username and password given to them on the computer in the room used.
* Information was provided about the home page of the website, basic topics, how to view the content, how to access it, and videos and games.
* It was explained that they should read the website for at least two hours a week, examine all sections and give feedback after two weeks.
* They were informed that they could contact the researcher 24/7 by e-mail and/or telephone if they had any problems regarding the website.
* This entire information process and filling out the data collection forms took 25 minutes.
* Two weeks after the first interview, the individuals included in the pre-application were administered the Website Analysis and Measurement Inventory Scale within the scope of the post-test at the Turkish Cypriot Diabetes Center.
* After the pre-application, the question "Do you have sufficient knowledge about diabetes?" in the "Socidemographic Questionnaire". and "Do you experience anxiety regarding insulin therapy?" The "I am undecided" option has been added to the questions. No changes were made to the scales.
* Individuals who were included in the preliminary application were not included in the scope of the research.
* After the research was completed, the username and passwords given for the preliminary application were cancelled. Individuals included in the pre-application were informed that the permanent address of the website would be sent to them via SMS.

Ethical Aspect of Research Necessary ethical permissions to conduct the research were obtained from Near East University and Turkish Cypriot Diabetes Association. In addition, for the use of scales in the research, Assoc. Prof. for the Diabetes Self-Care Activities Survey. Dr. From Gülhan Coşansudan, Prof. for the Diabetes-Specific Quality of Life Scale. Dr. Written consent was obtained from Ayşegül Kaptanoğlu, the researchers and the individuals participating in the research.

Limitations of the Research The scope of the research,

* Individuals who have internet connection at home or have internet on their mobile phone,
* Evaluation of only three-month effects,
* One of the limitations of the study is that it is based on self-report. Research Variables

Independent variables:

• Sociodemographic characteristics of the participants.

Dependent variables:

Participants;

* Quality of Life Specific to Diabetes,
* Diabetes Self-Care Activities Scale score averages.

Evaluation of Data The data will be evaluated in the SPSS 21.0 statistical program. Frequency and percentage analyzes will be performed for categorical variables, and mean and standard deviation analyzes will be performed for continuous variables.

In comparing the research variables, their suitability for normal distribution will be evaluated and then further statistical analyzes will be carried out. The research will be conducted with a 95% confidence interval and a 0.05% margin of error.

ELIGIBILITY:
Inclusion Criteria:• Turkish literate,

* Having access to the Internet,
* Diagnosed with Type II Diabetes,
* Mentally competent,
* Individuals who volunteered to participate in the study were recruited.

Exclusion Criteria:

* Cannot use a computer or smartphone,
* Under 18 years of age,
* Those with Type 1 Diabetes
* Working in the field of health and receiving health education in any field,
* Individuals who participated in the preliminary application were not included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Diabetes-Specific Quality of Life | 3 months
  It consists of four subscales, including diabetes-related anxiety and social/occupational anxiety, and 46 items. Each item in the scale is scored between 1-5 points. In the dimension of psychological satisfaction with the treatment (questions 22-24), the answer "very satisfied" is calculated as 1 point, the answer "very dissatisfied" is calculated as 5 points, while in other dimensions the answer "never" is calculated as 1 point, and the answer "always" is calculated as 5 points. The total score of the scale varies between 46-230. The total scale score and each subscale score are divided by the number of items, and the scores of 1 are converted into 5 points to obtain the total scale score. According to the scale total scores, high scores indicate good quality of life. The Turkish validity and reliability study of the scale was conducted by Yıldırım.
Diabetes Self-Care Activities | 3 months
  The Diabetes Self-Care Activities Questionnaire was developed by Toobert. In the survey, individuals; It is asked how many days (days/week) in the last seven days the patient performed self-care activities under the headings of diet, exercise, blood sugar test, foot care and smoking. The answers are marked as days (0-7) on a number line, and the 11th item, which only questions smoking, is stated as 0 - I do not smoke, 1 - I smoke (amount/piece of cigarettes smoked). Each subscale of the scale is scored separately and can be used independently.
  The Turkish validity and reliability study of the scale was conducted by Coşansu.

CONTACTS AND LOCATIONS:
Overall Officials: Kemal KE Elyeli, PhD(c)., Principal Investigator — Near East University
Locations (1):
- Near East University, Mersin, Lefkoşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No